CLINICAL TRIAL: NCT07121725
Title: Relationship of Dynamic Knee Valgus With Foot Posture, Pain, and Balance in Chronic Ankle Instability.
Acronym: DKV/CAI
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Meriam Nasser William Shafik, demonstrator of Musculoskeletal Disorders and it's Surgeries- Beni Suef University, Cairo University
Other Study IDs: No:P.T.REC/012/005728
Record Dates: First submitted 2025-08-03; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Ankle Instability
Keywords: Frontal plane projection angle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to identify if there is a relationship between the frontal plane projection angle as a measure of dynamic knee valgus with foot posture, pain, and dynamic balance in chronic ankle instability patients.

DETAILED DESCRIPTION:
The study design is an observational, correlational study to find if there is any relationship between the frontal plane projection angle with foot posture, pain, and dynamic balance in chronic ankle instability non-athletic patients.

The sample size is estimated to be 84. The frontal plane projection angle will be measured using a single-leg squat test and analyzed using Kinovea software.

Foot posture will be measured using the foot posture index. pain will be measured using a numerical rating scale. dynamic balance will be measured using modified star excursion balance tets

ELIGIBILITY:
Inclusion Criteria:

* A history of at least 1 significant ankle sprain.
* The initial sprain must have occurred at least 12 months prior to study enrollment.
* The most recent injury must have occurred more than 3 months prior.
* Additionally, a sprain that was associated with inflammatory symptoms (pain, swelling, etc.), Created at least 1 interrupted day of desired physical activity.
* A history of the previously injured ankle joint as "giving way" and/or recurrent sprain and/or "feelings of instability." And the self-reported outcome measure foot and ankle ability measure (FAAM): ADL scale <90%.

Exclusion Criteria:

* History of previous surgeries or fractures to the musculoskeletal structures (i.e., bones, joint structures, nerves) in either limb.
* No acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months, which impacted joint integrity and function (i.e., sprains, fractures) resulting in at least 1 interrupted day of desired physical activity.
* Participants were screened to exclude scoliosis using the Adam's Forward Bend Test (AFBT).

Ages: 15 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample will be recruited from the outpatient clinic of the Faculty of Physical Therapy at Cairo University by referral from the orthopedic doctor diagnosed with chronic ankle instability.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
correlation between the frontal plane projection angle and foot posture in chronic ankle instability patients. | baseline (single assessment session)
  NAME OF THE MEASUREMENT: "Frontal Plane Projection Angle"
  UNIT OF MEASURE: "measured in degrees"
  MEASUREMENT TOOL: "using a digital camera and Kinovea software"
  regarding foot posture:
  NAME OF THE MEASUREMENT: "Foot Posture"
  MEASUREMENT TOOL: "assessed using the Foot Posture Index (FPI), a 6-item scale" Criteria assessed included palpating the talar head, assessing supra and infra lateral malleolar curvature, calcaneal inversion/eversion, and examining talo-navicular prominence. Additionally, the congruence of the medial longitudinal arch and the forefoot's abduction/adduction relative to the rearfoot was evaluated
  UNIT OF MEASURE: "scored from -12 to +12
  * Highly supinated foot scores between (-5 to -12)
  * Supinated foot scores between (-4 to -1)
  * Normal foot scores between (0 to +5)
  * Pronated foot scores between (+6 to +9)
  * Highly pronated foot scores between (+10 to +12).
correlation between the frontal plane projection angle and pain in chronic ankle instability patients | baseline (single assessment session)
  regarding the frontal plane projection angle:
  NAME OF THE MEASUREMENT: "Frontal Plane Projection Angle"
  UNIT OF MEASURE: "measured in degrees"
  MEASUREMENT TOOL: "using a digital camera and Kinovea software"
  regarding pain measurement: NAME OF THE MEASUREMENT: Pain Intensity
  UNIT OF MEASURE:
  scale extending from 0 to 10 where 0 represented "no pain" and 10 represented the "worst pain possible''
  MEASUREMENT TOOL: 11-point Numeric Rating Scale (NRS-11)
correlation between the frontal plane projection angle and dynamic balance in chronic ankle instability patients. | baseline (single assessment session)
  regarding the frontal plane projection angle:
  NAME OF THE MEASUREMENT: "Frontal Plane Projection Angle"
  UNIT OF MEASURE: "measured in degrees"
  MEASUREMENT TOOL: "using a digital camera and Kinovea software"
  regarding dynamic balance:
  NAME OF THE MEASUREMENT: "Dynamic Balance"
  MEASUREMENT TOOL: "Modified Star Excursion Balance Test (M-SEBT)"
  UNIT OF MEASURE: "normalized reach distance in centimeters (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Meriam N Shafik, B.Sc, Principal Investigator — department of musculoskeletal disorders and it's surgery- Faculty of Physical Therapy
Locations (1):
- Faculty of Physical Therapy- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No